| Medi Stat<br>Statistics in Medicine | DOCUMENT NUMBER: 050-BST-PLN-001 | |
|---|---|---|
| TITLE: Statistical Analysis Plan of Protocol Number RZL-012-FD-P2aUS-001 | | EFFECTIVE DATE: 02/05/2019<br>REVISION NUMBER: 1.0 |

# **Revision History**

| Revision | <b>Revision Date</b> | Reason for Revision/Change Request | Revised By |
|---|---|---|---|
| 1.0 | 04-April-2019 | Original Release | Alexandra Perez-Alterman, |
| | | | Senior Biostatistician |
| 2.0 | 02-May-2019 | Update following Raziel.Ltd comments | Alexandra Perez-Alterman, |
| | | | Senior Biostatistician |
| 3.0 | 20-May-2019 | Update following Raziel.Ltd comments | Alexandra Perez-Alterman, |
| | | | Senior Biostatistician |

| Medi Stat<br>Statistics in Medicine | DOCUMENT NUMBER: 050-BST-PLN-001 | |
|---|---|---|
| TITLE: Statistical Analysis Plan of Protocol Number RZL-012-FD-P2aUS-001 | | EFFECTIVE DATE: 02/05/2019<br>REVISION NUMBER: 1.0 |

# Statistical Analysis Plan

An open label, phase 2a clinical trial for the evaluation of safety and efficacy of RZL-012 for the treatment of women with lipedema involving substantial fat above the knee or of women and men with nodular Dercum's disease

Protocol Number RZL-012-FD-P2aUS-001



DOCUMENT NUMBER: 050-BST-PLN-001


TITLE: Statistical Analysis Plan of Protocol Number RZL-012-FD-P2aUS-001

**EFFECTIVE DATE:** 02/05/2019 **REVISION NUMBER:** 1.0

# TABLE OF CONTENTS

| S | IGN A | ATURES PAGE | 4 |
|---|---|---|---|
| 1. | D | DEFINITIONS AND/OR ABBREVIATIONS | 5 |
| 2. | P | URPOSE | 9 |
| 3. | S | COPE | 9 |
| 4. | R | ESPONSIBILITies | 10 |
| | 4.1 | Medistat Ltd. Responsibilities | 10 |
| | 4.2 | Raziel Therapeutics's Responsibilities | 10 |
| 5. | P | ROCEDURE | 11 |
| | 5.1 | Introduction | 11 |
| | 5.2 | Rationale | 11 |
| | 5.3 | Study Objectives and Endpoints | 12 |
| | 5.4 | Overall study design and plan | 12 |
| | 5.5 | Selection of study population | 16 |
| | 5.6 | Statistical Analysis Software and Data Management | 16 |
| | 5.7 | Subject Population for analyses | 16 |
| | 5.8 | Statistical Analysis | 17 |
| 6. | R | ELATED DOCUMENTS (optional) | 19 |
| | 6.1 | Study Protocol: Protocol V7 - RZL-012-FD-P2aUS-001.7_CLEAN.docx | 19 |
| 7. | R | ELATED FORMS (optional) | 19 |
| 8. | R | EFERENCES | 19 |
| 9. | A | ppendices (optional) | 20 |
| | 9.1 | APPENDIX I: TABLE SHELLS | 20 |
| | 9 2 | APPENDIX II: LISTINGS SHELLS | 2322 |



| SIGNATURES PAGE | |
|-----------------------------------------|------------------|
| Alexandra Perez-Alterman, author | |
| Senior Biostatistician & SAS programmer | |
| MediStat Ltd. | Date: 11/06/1019 |
| JF | |
| David Israel | |
| Senior Biostatistician & SAS programmer | |
| MediStat Ltd. | Date: |
| Rachel Gueta | |
| Raziel Therapy Ltd. | Date: |

| Medi Stat<br>Statistics in Medicine | DOCUMENT NUMBER: 050-BST-PLN-001 | |
|---|---|---|
| TITLE: Statistical Analysis Plan | of Protocol Number RZL-012-FD-P2aUS-001 | EFFECTIVE DATE: 02/05/2019<br>REVISION NUMBER: 1.0 |

# 1. DEFINITIONS AND/OR ABBREVIATIONS

| Adverse event Alkaline phosphatase Alanine aminotransferase Aspartate aminotransferase Anatomical Therapeutic Chemical |
|---|
| Alanine aminotransferase Aspartate aminotransferase |
| Aspartate aminotransferase |
| Anatomical Therapeutic Chemical |
| · |
| Adenosine triphosphate |
| Area under the concentration-time curve |
| Brown-like adipose tissue |
| Body Mass Index |
| Blood urea nitrogen |
| Degrees Celsius |
| Complete blood count |
| Current Good Manufacturing Practices |
| Confidence Interval |
| Creatine Kinase - Muscle |
| Maximum observed concentration |
| Clinically not significant |
| Creatine phosphokinase |
| Case Report Form |
| Clinical Research Organization |
| C-reactive protein |

| Medi-Stat<br>Statistics in Medicine | DOCUMENT NUMBER: 050-BST-PLN-001 | |
|---|---|---|
| TITLE: Statistical Analysis Plan of Protocol Number RZL-012-FD-P2aUS-001 | | EFFECTIVE DATE: 02/05/2019<br>REVISION NUMBER: 1.0 |

| CTCAE | Common Terminology Criteria for Adverse Events |
|---|---|
| DLT | Dose-limiting toxicity |
| EC | Ethics Committee |
| ECG | Electrocardiogram |
| EF | Efficacy analysis set |
| FDA | Food and Drug Administration |
| FFA | Free fatty acids |
| FIFO | First In First Out |
| FOB | Functional Observational Battery |
| GLP | Good Laboratory Practice |
| GTTP | Gamma-glutamyltransferase |
| HbSAg | Hepatitis B surface antigen |
| HCV | Hepatitis C virus |
| HED | Human equivalent dose |
| HIV | Human immunodeficiency virus |
| IB | Investigator's Brochure |
| IC <sub>50</sub> | Half maximal inhibitory concentration |
| ICF | Informed Consent Form |
| ICH-GCP | International Conference on Harmonization Good Clinical Practice |
| IND | Investigational New Drug |
| INR | International normalized ratio |
| IRB | Institutional Review Board |
| LDL | Low-density lipoprotein |
| LDH | Lactate dehydrogenase |

| Medi-Stat<br>Statistics in Medicine | DOCUMENT NUMBER: 050-BST-PLN-001 | |
|---|---|---|
| TITLE: Statistical Analysis Plan of Protocol Number RZL-012-FD-P2aUS-001 | | EFFECTIVE DATE: 02/05/2019<br>REVISION NUMBER: 1.0 |

| LPL | Lipoprotein lipase |
|------------------|-----------------------------------------------|
| MEDDRA | Medical Dictionary for Regulatory Activities |
| MRI | Magnetic Resonance Imaging |
| NOAEL | No observed adverse effect level |
| NORD | National Organization for Rare Disorders |
| Pl | Principal Investigator |
| PK | Pharmacokinetics |
| PKA | PK Analysis set |
| PT | Prothrombin time |
| PTT | Partial thromboplastin time |
| QA | Quality Assurance |
| QOL | Quality of life |
| RBC | Red blood cells |
| RDW | Red cell distribution width |
| SA | Safety analysis set |
| SAE | Serious adverse event |
| SAP | Statistical Analysis Plan |
| SAS | Statistical Analysis Software |
| SAT | Subcutaneous adipose tissue |
| SC | Subcutaneous |
| SFM | Subcutaneous fat mass |
| SUSAR | Suspected Unexpected Serious Adverse Reaction |
| T <sub>1/2</sub> | Terminal half-life |
| TAG | Triacylglycerols |

| Medi Stat<br>Statistics in Medicine | DOCUMENT NUMBER: 050-BST-PLN-001 | |
|---|---|---|
| TITLE: Statistical Analysis Plan | of Protocol Number RZL-012-FD-P2aUS-001 | EFFECTIVE DATE: 02/05/2019<br>REVISION NUMBER: 1.0 |

| TG | Triglycerides |
|------------------|-----------------------------------------------|
| TLA | Tumescent Liposuction (Local Anesthesia) |
| T <sub>max</sub> | Time of maximum observed sample concentration |
| UCP1 | Uncoupling protein 1 |
| US/USA | United States/United States of America |
| WAL | Water Assisted Liposuction |
| WAT | White adipose tissue |
| WBC | White blood cells |
| WHO | World health organization |

| Medi Stat<br>Statistics in Medicine | DOCUMENT NUMBER: 050-BST-PLN-001 | |
|---|---|---|
| TITLE: Statistical Analysis Plan of Protocol Number RZL-012-FD-P2aUS-001 | | EFFECTIVE DATE: 02/05/2019<br>REVISION NUMBER: 1.0 |

## 2. PURPOSE

- 2.1 The purpose of this document is to describe in detail the Statistical Analysis Plan of clinical study procedures carried out by Medistat Ltd.
- 2.2 This document serves Medistat Ltd. as a guiding document for all statistical analyses performed at the end of each clinical study.
- 2.3 This SAP is specific to Raziel Therapeutics Ltd., study RZL-012-FD-P2aUS-001.
- 2.4 This SAP aims to provide details on: sample size calculation, efficacy analyses and safety analyses.

## 3. SCOPE

- 3.1 This document applies to all members of the statistical & data management units in Medistat Ltd.
- 3.2 This document includes the main and interim study trial analysis.

| Medi Stat<br>Statistics in Medicine | DOCUMENT NUMBER: 050-BST-PLN-001 | |
|---|---|---|
| TITLE: Statistical Analysis Plan of Protocol Number RZL-012-FD-P2aUS-001 | | EFFECTIVE DATE: 02/05/2019<br>REVISION NUMBER: 1.0 |

## 4. RESPONSIBILITIES

# 4.1 Medistat Ltd. Responsibilities

The following personnel are responsible for these activities:

| Activities | Responsible and | Title |
|---|---|---|
| | accountable | |
| Statistical Analysis Plan | Alexandra Perez-Alterman | Senior Biostatistician |
| (SAP) | | & SAS Programmer |
| Statistical Report and listing | Alexandra Perez-Alterman | Senior Biostatistician |
| appendix | | & SAS Programmer |
| Quality Assurance (QA) of | David Israel | Senior Biostatistician |
| SAP and programs | | & SAS Programmer |
| Quality Assurance (QA) of | Shimrit Herbst | Quality & Data |
| final report | | Assurance Manager |

# 4.2 Raziel Therapeutics's Responsibilities

- 4.2.1 To review and approve the SAP and related documents prior to database lock.
- 4.2.2 To review and approve the draft and final statistical report and listing appendix.

| Medi Stat<br>Statistics in Medicine | DOCUMENT NUMBER: 050-BST-PLN-001 | |
|---|---|---|
| TITLE: Statistical Analysis Plan of Protocol Number RZL-012-FD-P2aUS-001 | | EFFECTIVE DATE: 02/05/2019<br>REVISION NUMBER: 1.0 |

#### 5. PROCEDURE

#### 5.1 Introduction

- 5.1.1 This Statistical Analysis Plan (SAP) is based on the study protocol version 7, dated 03 January, 2019.
- 5.1.2 This Statistical Analysis Plan (SAP) contains details of the statistical analyses that will be performed, providing a more detailed description of the approach defined in the study protocol. Definitions of variables and populations used for the analyses are also included. The SAP will be finalized and signed prior to hard lock of the database.
- 5.1.3 General output specifications are provided; examples are given of calculations of derived variables.

#### 5.2 Rationale

- 5.2.1 The initial dose was determined by the NOAEL established by the Good Laboratory Practice (GLP) extended single dose toxicology study and by the previous phase 0 clinical trial in which 20mg RZL-012 was the highest dose achieved. This initial study is an escalating dose study. If no more than 1 subject experiences intolerable side effects within 14 days following the injection of the last dosed group, according to schedule, an additional cohort of volunteers will be administrated the next dose level.
- 5.2.2 Cohort 1- will be comprised of subjects with Dercum's disease. All subjects will be injected with RZL-012. Dosing will be calculated according to the size of the nodule (diameter) as determined by ultrasound: 5mg/cm2 reaching a maximal dose of 40 mg RZL-012 per subject (1/6.25 the NOAEL based on the Human Dose Equivalent [HED] GLP Toxicology studies).
- 5.2.3 Cohort 2 will be comprised of subjects with lipedema with substantial fat above the knee and will be conducted in a dose escalation manner.
- 5.2.4 The first 3 subjects will receive 60mg RZL-012 (1/4.688th the NOAEL based on HED from GLP toxicology study).
- 5.2.5 The last 3 subjects will receive 80mg RZL-012 (1/3.125th the NOAEL based on HED from GLP toxicology study).

| Medi Stat<br>Statistics in Medicine | DOCUMENT NUMBER: 050-BST-PLN-001 | |
|---|---|---|
| TITLE: Statistical Analysis Plan of Protocol Number RZL-012-FD-P2aUS-001 | | EFFECTIVE DATE: 02/05/2019<br>REVISION NUMBER: 1.0 |

- 5.3 Study Objectives and Endpoints
  - 5.3.1 Primary Objective
- 5.3.1.1 The primary endpoint will be the evaluation of the overall safety of RZL-012 injection into the subcutaneous fat in Dercum's disease and lipedema. The trial will proceed within a cohort provided that no more than one subject experiences intolerable side effects in a cohort.
  - 5.3.2 Secondary Objective
- 5.3.2.1 For lipedema subjects The reduction in local subcutaneous fat in the injection site region as compared to baseline as assessed by leg circumference above the knee assessments and by the reduction in nodules size and/or numbers assessed by ultrasound.
- 5.3.2.2 For Dercum's disease subjects The reduction in local subcutaneous fat in the injection site region as compared to baseline assessed by the reduction in nodules size and/or numbers by ultrasound.
- 5.3.2.3 Extended duration of the fat reduction effect. To that end, ultrasound images and circumference measurement will be followed for 56 days.
- 5.3.2.4 Elucidation of the tissue changes by ultrasound of the injection site to include reduction in fat thickness and nodular quality.
- 5.3.2.5 Improvement in local pain as measured by Comparative Pain Scale and by the reduction in the use of analgesics.
- 5.3.2.6 Improvement in QOL and function in lipedema subjects as measured by questionnaire (such as The Lower Extremity Functional Scale (LEFS)).
- 5.4 Overall study design and plan
  - 5.4.1 Study Design
- 5.4.1.1 Six subjects in cohort 1, all assigned to the RZL-012 treatment group will be dosed at a maximal dose of 40 mg RZL-012 (approximately 1/6.25th the NOAEL as determined in the GLP toxicology study). Dosing will be calculated according to the size of the nodule (diameter) as determined by ultrasound in a dose of 5mg/cm2:
- 5.4.1.2 Six subjects in cohort 2, all assigned to the RZL-012 treatment group, will be dosed as follows:



- 5.4.1.3 The first 3 subjects will receive 30mg RZL-012 in 6 injections (0.1mL each) in one leg followed by 30mg RZL-012 (6 injections, 0.1mL each) in the second leg adding up to 12 injections of 60mg RZL-012 (1/4.688th the NOAEL based on HED from GLP toxicology study).
- 5.4.1.4 The last 3 subjects will receive 40mg RZL-012 in 8 injections (0.1mL each) in one leg followed by 40mg RZL-012 (8 injections, 0.1mL each) in the second leg adding up to 16 injections of 80mg RZL-012 (1/3.125th the NOAEL based on HED from GLP toxicology study).
- 5.4.1.5 Dosing of subjects in each cohort will progress consecutively from one individual to the other at 7-day intervals. This study design will allow the physicians to monitor safety for at least 7 days prior to dosing the next subject. For cohort 2 the decision to proceed to the next dose level will be made after reviewing all safety data collected by Day 14 within  $2 \pm 1d$  of the last dosed subject. The trial will proceed within a cohort provided that no more than one subject experiences intolerable side effects in a cohort, and based on the decision made by the Principal Investigator (PI) and the Medical Monitor.

#### 5.4.2 Schedule of Assessments

| Study Procedure | Screening Day | Baseline<br>(Treatm<br>ent) | | v | isit Scheo | dule (Da | ys 1 to 2 | 8) | Follow-<br>up |
|---|---|---|---|---|---|---|---|---|---|
| Study Day <sup>a</sup> | Day <sup>a</sup> -(-14)<br>through Day<br>(-2) | Day <sup>a</sup> 0 | Day<br>1 | Day<br>3 | Day 7 | Day<br>14 | Day<br>21 | Day<br>28 | Day 56 |
| Signed informed consent | X | | | | | | | | |
| Medical history | X | | | | | | | | |
| Concomitant Medication | X | | | | | | | | |
| Complete physical exam | X | | | | | | | X | |
| Pain measurement | X | | | | | X | | X | X |
| For lipedema subjects - QOL measurement | X | | | | | X | | X | X |

| Medi Stat<br>Statistics in Medicine | DOCUMENT NUMBER: 050-BST-PLN-001 | |
|---|---|---|
| TITLE: Statistical Analysis Plan of Protocol Number RZL-012-FD-P2aUS-001 | | EFFECTIVE DATE: 02/05/2019 REVISION NUMBER: 1.0 |

| Serology assays (HbSAg, HCV, HIV) | X | | | | |
|---|---|---|---|---|---|
| Urine Drug Screen | X | | | | |
| Height and weight | X | | | | |
| For Dercum's disease<br>subjects – ultrasound<br>assessing nodules size<br>(diameter) and quality | X | | | | |
| For lipedema subjects – assessing fat thickness and nodular quality by ultrasound. | X | | | | |
| For lipedema subjects – measurement of leg circumference above the knee | X | Pre ° X | | | |
| For lipedema subjects – ultrasound assessing nodules to be injected For Dercum's disease subjects – ultrasound re- assessing nodules size | | Pre ° X | | | |
| Photography of site of injection | X | | X | | X |
| Serum Chemistry,<br>Hematology <sup>b</sup> | X | Pre <sup>c</sup> X | X | X | X |
| Urinalysis | X | | | | |
| Draize score at the injected site <sup>d</sup> | X | Pre <sup>c</sup> X post <sup>c</sup> | X | | X |

| Medi Stat<br>Statistics in Medicine | DOCUMENT NUMBER: 050-BST-PLN-001 | |
|---|---|---|
| TITLE: Statistical Analysis Plan of Protocol Number RZL-012-FD-P2aUS-001 | | EFFECTIVE DATE: 02/05/2019<br>REVISION NUMBER: 1.0 |

- a. Study day is based on Day 0 defined as the day of RZL-012 injection.
- CBC, coagulation, serum chemistry analysis, renal and liver function, urinalysis, CPK, amylase measurement: before injection,14d and 28d following injection
- c. Pre/post refers to before/after injection respectively
- d. Draize score evaluation: before injection, 2h, 24h and 7d, 14d, 21d and 28d following injection
- e. Vital signs measurement: before injection, 2h, 24h and 7d, 14d, 21d and 28d following injection
- f. ECG is to be performed in triplicate for all measurements in given time point: 4h, 8h, 24h following injection
- g. Pulse rate measurements at given time points: 1h, 2h, 4h, 8h, 24h following injection in the opposite hand of blood sampling

| Vital signs <sup>e</sup> | X | Pre <sup>c</sup> X | X | | X |
|---|---|---|---|---|---|
| Injection of RZL-012 | | X | | | |
| ECG <sup>f</sup> | X | X post c | X | | |
| Pulse rate <sup>g</sup> | | X post <sup>c</sup> | X | | |
| Subjects diary recording of analgesics use | X | X | X | X | X |
| AE assessment | | | X | ·<br> | |

| Medi Stat<br>Statistics in Medicine | DOCUMENT NUMBER: 050-BST-PLN-001 | |
|---|---|---|
| TITLE: Statistical Analysis Plan of Protocol Number RZL-012-FD-P2aUS-001 | | EFFECTIVE DATE: 02/05/2019<br>REVISION NUMBER: 1.0 |

- 5.4.3 Randomization, Blinding and Un-blinding
- 5.4.3.1 This is an open label study where all subjects will receive the investigational drug (RZL-012).
- 5.5 Selection of study population
  - 5.5.1 Study Population
- 5.5.1.1 Post-menopausal women no more than 65 years old, with lipedema involving substantial fat above the knee or nodular Dercum's disease in such women and in men 20- 65 years with nodular Dercum's disease.
  - 5.5.2 Rationale Sample Size Calculation
- 5.5.2.1 This study is planned following a 6 subjects per group paradigm. A maximum of 12 evaluable subjects will be included in the study (6 subjects with Dercum's disease and 6 subjects with lipedema) and followed for as long as 2 months.
- 5.6 Statistical Analysis Software and Data Management
  - 5.6.1 Data manipulation, tabulation of descriptive statistics, calculation of inferential statistics, and graphical representations will be performed using SAS® version 9.3 or higher for Windows. If the use of other software is warranted, the final statistical methodology report will detail what software was used for what purposes.
  - 5.6.2 Data Management
  - 5.6.3 Data management for the study is performed by Medistat.
  - 5.6.4 Medical Coding
  - 5.6.5 Concomitant medications entered into the database are coded using the WHO (World Health Organization) Drug Public Website Dictionary named WHOCC-ATC/DDD index, which employs the Anatomical Therapeutic Chemical classification system.
  - 5.6.6 Adverse events are coded using the most updated version of Medical Dictionary for Regulatory Activities (MedDRA) terminology.
  - 5.6.7 Medical history events are coded using the most updated version of Medical Dictionary for Regulatory Activities (MedDRA) terminology
  - 5.6.8 Handling of Missing data
  - 5.6.9 No imputation of missing data will be performed
- 5.7 Subject Population for analyses



- 5.7.1 The SA will consist of all enrolled subjects who received the study treatment, (exposed population), including subjects prematurely withdrawn.
- 5.7.2 All enrolled subjects receiving at least one study drug injection are considered evaluable for the SA set. The SA analysis set will serve as the principal data analysis set for the analyses of the safety endpoints.
- 5.7.3 The EF will consist of all subjects from the SA analysis set without any major protocol violations measured at baseline. Subjects will be analyzed according to the treatment received.
- 5.7.4 The SA analysis set will serve as the principal data analysis set for the analyses of the safety endpoints.
- 5.7.5 The EF analysis set will serve as the principal data analysis set for the analyses of the efficacy endpoints.

#### 5.8 Statistical Analysis

- 5.8.1 General
- 5.8.2 Statistical analyses will be mainly descriptive in nature where study data will be tabulated and summarized using the mean, standard deviation or standard error, median, minimum, maximum and number of subjects by cohort for continuous data. For categorical data, results will be summarized via a count and percentage by cohort. The results will be presented overall, per cohort and per cohort and dose. The effects of noncompliance, dropouts, and covariates, may be assessed to determine the impact on the general applicability of results from this study.
- 5.8.3 If any statistical tests are performed, they will be two-sided. The required significance level of findings will be equal to or lower than 5%. Nominal p-values will be presented.
- 5.8.4 Where confidence limits are appropriate, the confidence level will be 95%.
- 5.8.5 The data is analyzed using the SAS ® version 9.3 or higher (SAS Institute, Cary North Carolina).
- 5.8.6 Statistical methods presented in the SAP may be slightly different from those that are presented in the protocol. Differences are clearly stated and the SAP supersedes the protocol only with regard to the way data will be handled and analysed.



- 5.8.7 Subject Disposition
- 5.8.8 A detailed description of subject accountability including count of subjects included, exposed, completed (i.e., subjects who complete the study treatment) and discontinued along with the main reason for discontinuation will be generated for each cohort and for all subjects. All withdrawals from the study, taking place on or after study drug injection, will be fully documented in the body of the Clinical Study Report.
- 5.8.9 Note that the actual study duration is for a period of maximum 2 months, with efficacy analyses being conducted at 28 days and 56 days.
- 5.8.10 Demographic and Baseline Characteristics
- 5.8.11 Baseline will be defined as the last available and evaluable parameter value before and closest to the injection. If a rechecked value is used for baseline, it should be collected under the same conditions as for the planned baseline.
- 5.8.12 Baseline safety data will be presented along with subsequent safety values assessed during or after dosing.
- 5.8.13 The incidence of intolerable side effects will be presented overall and by cohort along with two sided 95% exact binomial Confidence Interval (CI).
- 5.8.14 Percent changes from baseline in local fat reduction (circumference of the leg above the knee, nodules size and/or numbers in the injected area) and tissue changes (fat thickness), will be presented in tabular form by visit.
- 5.8.15 Changes in nodular quality, local pain, quality of life and function will be presented in tabular form by visit and cohort.
- 5.8.16 Safety and Tolerability
- 5.8.17 Safety analyses will be descriptive in nature.
- 5.8.18 All reported AEs will be coded to a standard set of terms using MedDRA coding dictionary (V22.0 or higher) treatment.



- 5.8.19 AEs and tolerability data will be presented descriptively by treatment and cohort. AEs will be tabulated by body system, preferred term, seriousness, severity and relation to study drug by cohort. Where applicable, changes in values over time (e.g., lab values, vital signs, ECGs) will be presented; this will include clinical laboratory evaluations (including CBC, blood chemistry and urinalysis), coagulation (INR, PTT and PT), cytokines, vital signs, and ECGs. Shift tables of normal / abnormal versus baseline may be presented as well.
- 5.8.20 Draize scores will be presented in tabular format by visit, treatment, and cohort.
- 5.8.21 Concomitant medication verbatim terms (as recorded on the CRFs) will be coded to Anatomical Therapeutic Chemical (ATC) Level 2 and 4 using the World Health Organization (WHO) dictionary.

## 6. RELATED DOCUMENTS (OPTIONAL)

6.1 Study Protocol: Protocol V7 - RZL-012-FD-P2aUS-001.7 CLEAN.docx

## 7. RELATED FORMS (OPTIONAL)

Not Applicable

#### 8. REFERENCES

Not Applicable

| MediStat Statistics in Medicine | DOCUMENT NUMBER: 050-BST-PLN-001 | |
|---|---|---|
| TITLE: Statistical Analysis Plan of Protocol Number RZL-012-FD-P2aUS-001 | | EFFECTIVE DATE: 02/05/2019<br>REVISION NUMBER: 1.0 |

## 9. APPENDICES (OPTIONAL)

9.1 APPENDIX I: TABLE SHELLS

14.1 Demographic Data

Table 14.1-1: Disposition of Subjects

Table 14.1-2: Analysis populations

Table 14.1-3: Demographic Data (Part 1 of 2)

Table 14.1-3: Demographic Data (Part 2 of 2)

Table 14.1-4: Medical History

Table 14.1-5: Disease-Related Medical History

14.1-6: Disease characteristics

Table 14.1-6-1: Dercum's cohort lipoma type

Table 14.1-6-2: Lipedema disease characteristics (Part 1 of 2)

Table 14.1-6-2: Lipedema disease characteristics (Part 2 of 2)

14.2 Drug administration

Table 14.2-1 Drug administration

14.3 Efficacy Assessment

Table 14.3-1 Pain by comparative scale by cohort

Table 14.3-2 Reduction in Pain from baseline by visit

Table 14.3-3 Relative Change in local pain

14.3-4 Dercum's disease cohort

Table 14.3-4-1 Number of Lipomas by visit

Table 14.3-4-2 Reduction of number of Lipomas from baseline by visit

Table 14.3-4-3 Relative Change in Number of lipomas

Table 14.3-4-4 Size of lipomas by visit and type

| Medi Stat<br>Statistics in Medicine | DOCUMENT NUMBER: 050-BST-PLN-001 | |
|---|---|---|
| TITLE: Statistical Analysis Plan of Protocol Number RZL-012-FD-P2aUS-001 | | EFFECTIVE DATE: 02/05/2019<br>REVISION NUMBER: 1.0 |

Table 14.3-4-5 Reduction\*\* in Size of lipomas by visit and type

Table 14.3-4-6 Relative change in Size of lipomas by visit and type

Table 14.3-4-7 Lipoma description

14.3-4.8 Correlation between pain and size of lipomas

Table 14.3-4.8-1 Correlation between lipoma size and pain for lipomas with Fibrotic tissue not associated with the capsule

Table 14.3-4.8-2 Correlation between lipoma size and pain for lipomas with Fibrotic tissue associated with the capsule

Table 14.3-4.8-3 Correlation between reduction in lipoma size and reduction in pain for all lipomas

# 14.3-5 Lipedema cohort

Table 14.3-5-1 Number of fat locations by visit

Table 14.3-5-2 Thickness of fat locations by visit for right/left leg

Table 14.3-5-3 Reduction\*\* in fat locations Thickness by visit and type

Table 14.3-5-4 Relative change in fat locations Thickness by visit and type

Table 14.3-5-5 Fat tissue description

Table 14.3-5-6 Nodule description

Table 14.3-5.7 Correlation between reduction in nodule size and reduction in pain

Table 14.3-5-8 Additional measurements

Table 14.3-5-9 Reduction\*\* in additional measurements

Table 14.3-5-10 Relative change in additional measurements

## 14.4 Safety Data and Other Assessments

#### 14.4.1 Adverse Events

Table 14.4.1-1: Frequency of Any Adverse Events



Table 14.4.1-2: Frequency of any intolerable side effects

Table 14.4.1-3: Summary of Adverse Events by SOC and PT by treatment

Table 14.4.1-4: Summary of Adverse Events by SOC, PT, severity and by treatment

Table 14.4.1-5: Summary of Adverse Events by SOC, PT, relationship to study treatment and by treatment

#### 14.4.2 Other Assessments

Table 14.4.2-1: Summary of Vital signs

Table 14.4-2.2 Changes in Vital signs

Table 14.4-2.3 Relative Changes in Vital signs

Table 14.4-2.4: Laboratory tests

Table 14.4-2.5: Draize Score

Table 14.2-3.6 ECG results

Table 14.2-3.7 Changes in ECG results

Table 14.2-3.8 Relative Changes in ECG results

| Medi Stat<br>Statistics in Medicine | DOCUMENT NUMBER: 050-BST-PLN-001 | |
|---|---|---|
| TITLE: Statistical Analysis Plan of Protocol Number RZL-012-FD-P2aUS-001 | | EFFECTIVE DATE: 02/05/2019<br>REVISION NUMBER: 1.0 |

#### 9.2 APPENDIX II: LISTINGS SHELLS

16.2.1 Subject Disposition

Listing 16.2.1-1: Subject Disposition

Listing 16.2.1-2: Visit dates per subject

Listing 16.2.1-3: Unscheduled Visit

16.2.2 Protocol Deviations

Listing 16.2.2-1: Inclusion/Exclusion criteria violations

16.2.3 Demographic Data and Baseline Assessments

Listing 16.2.3-1: Demographic Data

Listing 16.2.3-2: Medical History

Listing 16.2.3-3: Disease-Related Medical History

16.2.3-4: Disease characteristics

Listing 16.2.3-4-1: Dercum's disease cohort lipoma type

Listing 16.2.3-4-2: Lipedema cohort disease characteristics

16.2.4 Compliance/Exposure/Drug Concentration Data

Listing 16.2.4-1: Injection of RZL-012 (Part 1 of 2)

Listing 16.2.4-1: Injection of RZL-012 (Part 2 of 2)

16.2.5 Individual Efficacy/Response Data

Listing 16.2.5-1: Comparative pain for both cohort

16.2.5-2 Ultrasound and measurements Dercum's cohort

Listing 16.2.5-2-1: Number of Lipomas

Listing 16.2.5-2-2: Lipomas description

Listing 16.2.5-2-3: Size of Lipomas

16.2.5-3 Ultrasound and measurements Lipedema cohort

Listing 16.2.5-3-1: Number of Injected Fat Locations

Listing 16.2.5-3-2: Fat tissue description

Listing 16.2.5-3-3: Fat tissue description

Listing 16.2.5-3-4: Thickness of Fat Tissue

Listing 16.2.5-3-5: Thickness of Fat Tissue - Shift table

Listing 16.2.5-3-6: Average reduction in Thickness of Fat Tissue



Listing 16.2.5-3-7: Additional measurements

Listing 16.2.5-3-8: Additional measurements - Shift table

16.2.6 Adverse Events listings

Listing 16.2.6-1: All Adverse events (Part 1 of 2)

Listing 16.2.6-1: Adverse events (Part 2 of 2)

Listing 16.2.6-2: Serious Adverse Events (Part 1 of 2)

Listing 16.2.6-2: Serious Adverse Events (Part 2 of 2)

16.2.7 Laboratory and other safety parameters

Listing 16.2.7-1: Laboratory tests (Part1 of 2)

Listing 16.2.7-1: Laboratory tests (Part 2 of 2)

Listing 16.2.7-2: ECG Results\* (Part 1 of 2)

Listing 16.2.7-2: ECG Results\* (Part 2 of 2)

Listing 16.2.7-3: Vital signs (Part 1 of 2)

Listing 16.2.7-3: Vital signs (part 2 of 2)

Listing 16.2.7-4: Draize Score

Listing 16.2.7-5: Benadryl

Listing 16.2.7-6: Concomitant Medications (Part 1 of 3)

Listing 16.2.7-6: Concomitant Medications (Part 2 of 3)

Listing 16.2.7-6: Concomitant Medications (Part 3 of 3)

Listing 16.2.7-7: Comments